CLINICAL TRIAL: NCT04025619
Title: Development of Novel Adhesive Sports Tape Modular to Facilitate Use of Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Juin-Hong Cherng, Assistant Professor, National Defense Medical Center, Taiwan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GreenE2017
Record Dates: First submitted 2017-12-18; First posted 2019-07-19 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: 2 groups of participant, one of the group took the questionnaire then received the intervention for seven days, then took the same questionnaire again.
  The other group took the physical examination and received the intervention immediately, then took the physical examination again when the intervention is on the treating area.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): the data is collected from the same participant after the intervention.
  Interventions: Device: tape
- Control group (No Intervention): The Collect the data from the same participant before the intervention as control

INTERVENTIONS:
Device: tape — Sports tape
  Arms: treatment group

SUMMARY:
Special metals (e.g. Germanium, Titanium, and π element) can be used to produce far-infrared radiation. The applications of these metals in promoting blood circulation are worth investigating. This clinical trial recruited subjects for using tape made up of Ge, Ti, and π element developed by Green Energy Nano Technology Co., Ltd. We assumed that the experimental tape can improve the participants' peripheral blood circulation and their quality of life. In this clinical trial, the clinical efficacy and safety of the test products were assessed using physical examination and questionnaires.

DETAILED DESCRIPTION:
This study is made of two open-labeled, two-arm studies. 20 to 80 years old patient diagnosed with varicose veins were included in the study. Besides, patient with the following characteristics was excluded: vulnerable group, patient with an open wound at lower limb which cannot be taped, unable to express willingness clearly, Dyslexia, and inability to ambulate.

The final number of total participant is 86 participants and 66 out of 86 participants were assigned to the first study which is divided into 2 groups, the experimental and control group. The experimental group received the experimental tape as treatment, and the control group didn't receive any treatment. The participants will fill in the questionnaires including visual Analogue Scale and quality of life on the first day of the study, and fill the same questionnaires seven days later.

Furthermore, the rest of the 20 participants were assigned to the second study. The researchers evaluate their peripheral blood circulation by Segmental Blood Pressure over Pulse Volume Recording (SBP/PVR), Maximum Venous Outflow over Segmental Venous Capacitance (MVO/SVC), and Ankle Brachial Index (ABI) before they received the treatment, then the researchers inspect the same indexes after they received the treatment right after the first tests.

ELIGIBILITY:
Inclusion Criteria:

* Cardiovascular disease (deep Vein Thrombosis or Chronic venous insufficiency)

Exclusion Criteria:

* Vulnerable populations
* wound at lower limb which can not take the intervention
* one can not make express consent clearly
* dyslexia
* who need physical assistance during ambulation
* nonfunctional ambulator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Ankle-Brachial Pressure Index | 1 day
  Detect the pressure difference in percentage between brachial pressure and ankle pressure by the pulse volume record and ultrasound device.
MVO/SVC | 1 day
  The ratio of maximum venous outflow (MVO) to the segmental venous capacitance (SVC)
Visual Analog Scale (VAS) Pain | 1 day
  VAS is measurement instrument for describing pain severity or intensity. The pain scale is range from 0 to 10, representing "no hurt" to "hurt worst", respectively.

SECONDARY OUTCOMES:
Kidney Disease Quality of Life | Day 0 (before intervention) and Day 7 (after using the intervention for 7 days)
  Questionnaire to assess generic and kidney-disease targeted aspects of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- National Defense of Medical Center, Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No